CLINICAL TRIAL: NCT00073593
Title: A Study Comparing Angiomax (Bivalirudin) to Heparin With Protamine Reversal in Patients Undergoing Coronary Artery Bypass (OPCAB) Surgery
Brief Title: Comparing Angiomax to Heparin With Protamine Reversal in Patients OPCAB
Acronym: OPCAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-02-07; EVOLUTION
Record Dates: First submitted 2003-11-26; First posted 2003-11-27 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass Surgery
Keywords: Off-Pump Coronary Artery Bypass Graft Surgery; CABG; OPCAB; Heparin; Patients requiring off-pump CABG
MeSH Terms: interventions — bivalirudin; Heparin; Protamines

ARMS (2):
- bivalirudin (Experimental): 250mg vial given as 0.75mg/kg intravenous (IV) bolus and 1.75 mg/kg/hr IV infusion for the duration of the procedure with the option to increase or decrease the infusion in 0.25 mg/kg/hr increments or to administer additional 0.1-0.5 mg/kg boluses to maintain an ACT>300 seconds.
  Interventions: Drug: Bivalirudin
- heparin/protamine (Active Comparator): 1.5-3.5 mg/kg (200-400 U/kg) intravenous (IV) bolus to target an ACT >300 seconds followed by weight-adjusted boluses as needed during the procedure to achieve/maintain the target ACT. Protamine as needed
  Interventions: Drug: Heparin; Drug: Protamine

INTERVENTIONS:
Drug: Bivalirudin — 250 mg vial administered as 0.75 mg/kg intravenous (IV) bolus and 1.75 mg/kg/h IV infusion for the duration of surgery with the option to increase or decrease the infusion in 0.25 mg/kg/h increments or to administer additional 0.1-0.5 mg/kg boluses to maintain an activated clotting time (ACT) >300 seconds (s).
  Arms: bivalirudin
Drug: Heparin — : Per institutional practice, at 1.5-3.5 mg/kg (200-400 U/kg) IV bolus to achieve a target ACT of >300 s followed by weight-adjusted boluses as needed during surgery to achieve/maintain the target ACT. Batches from hospital stock.
  Arms: heparin/protamine
Drug: Protamine — Per institutional practice. Batches from hospital stock.
  Arms: heparin/protamine

SUMMARY:
The purpose of this study is to examine the safety and efficacy of Angiomax as an alternative anticoagulant to heparin with protamine reversal in patients undergoing off-pump coronary artery bypass graft surgery.

ELIGIBILITY:
Inclusion:

* Provide written informed consent before initiation of any study related procedures.
* Be at least 18 years of age.
* Be accepted for elective off-pump coronary artery bypass graft (CABG) surgery without concomitant cardiac surgical procedures.
* < 4 planned Coronary Artery Bypass Grafts

Exclusion:

* Any prior Cardio-Thoracic Surgical procedures requiring median sternotomy
* Confirmed pregnancy - baseline urine or serum pregnancy test (if woman of childbearing potential).
* Cerebrovascular accident within 6 months before randomization, or any cerebrovascular accident with residual neurological deficit.
* Intracranial neoplasm, arteriovenous malformation, or aneurysm.
* Dependency on renal dialysis or creatinine clearance <30mL/min.
* Ongoing treatment with warfarin (or other oral anticoagulants) at the time of randomization. Patients previously treated with warfarin may be enrolled if warfarin therapy can be safely discontinued and baseline INR is <1.3 times control in the absence of heparin therapy.
* Known allergy to Angiomax or hirudin derived drugs, or known sensitivity to any component of these products.
* Patients receiving clopidogrel within the previous 5 days of randomization.
* Patients receiving a glycoprotein IIb/IIIa inhibitor within 48 hours if abciximab (ReoPro) or within 24 hours if eptifibatide (Integrilin) and tirofiban (Aggrastat) of randomization
* Patients receiving lepirudin or argatroban within the previous 24 hours of randomization.
* Patients receiving low molecular weight heparin (LMWH) or thrombolytics within the previous 12 hours or unfractionated heparin within 30 minutes of randomization.
* Patients with active or prior history of heparin-induced thrombocytopenia (HIT)/heparin-induced thrombocytopenia and thrombosis syndrome (HITTS)*.
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of randomization.
* Refusal to undergo blood transfusion should it become necessary.
* Any other disease or condition, which, in the judgment of the investigator would place a patient at undue risk by being enrolled in the trial or inability to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-08; Primary Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Death | Hospital discharge or Day 7
Q-wave MI | hospital discharge or day 7,
Repeat Coronary Revascularization, | hospital discharge or day 7,
Stroke (hemorrhagic or ischemic). | hospital discharge or day 7

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sternlicht, MD, Study Director — The Medicines Company
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States